CLINICAL TRIAL: NCT01742039
Title: A New Therapeutic Strategy to Reduce the Incidence of Postoperative Atrial Fibrillation
Brief Title: Prevention of Postoperative Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Other Study IDs: AF01
Record Dates: First submitted 2012-11-14; First posted 2012-12-05 (Estimated); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Postoperative Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- b-blocker
- amiodarone
- atrial pacing
- amiodarone plus atrial pacing

SUMMARY:
The primary aim of this study is to determine the safest and most effective therapeutic strategy to decrease the incidence of postoperative atrial fibrillation following cardiac surgery in an era with shorter ICU and hospital length of stay. A secondary goal is to evaluate the length of hospital stay associated with each treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* age > or = to 18 years
* sinus rhythm
* undergoing either coronary artery bypass graft surgery (CABG), valvular heart surgery or a combined procedure

Exclusion Criteria:

* received a class-I or class-III antiarrhythmic agent in the past six months
* had second or third degree heart block
* had a resting heart rate of less than 50 beats per minute
* had a systolic blood pressure less than 100 mmHg
* had severe asthma or severe chronic obstructive pulmonary disease
* had uncontrolled heart failure
* had a serum aspartate aminotransferase or alanine aminotransferase concentration greater than four times the upper limit of normal

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patients undergoing open heart surgery
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2008-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
occurrence of atrial fibrillation | postoperative day 0-day of discharge (an average of 5 days)
  The primary endpoint of this study was also the occurrence of atrial fibrillation for any length of time requiring treatment as a result of symptoms or hemodynamic compromise.
occurrence of atrial fibrillation | postoperative day 0-day of discharge (an average of 5 days)
  The primary endpoint of this study was the occurrence of atrial fibrillation lasting longer than five minutes

SECONDARY OUTCOMES:
length of stay | participants will be followed for the duration of hospital stay, an expected average of 5 days
  The secondary endpoint was the length of hospital stay after surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - George Washington University Hospital, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia